CLINICAL TRIAL: NCT00122057
Title: Impact of Antibiotic Treatment on Outcome in Patients With Ventilator-Associated Tracheobronchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: University Hospital, Lille, University Hospital, Lille
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005/0506
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2006-09

CONDITIONS: Respiratory Tract Diseases; Nosocomial Infections
Keywords: ventilator-associated tracheobronchitis; nosocomial tracheobronchitis
MeSH Terms: conditions — Respiratory Tract Diseases; Cross Infection

INTERVENTIONS:
Drug: antibiotic treatment

SUMMARY:
The aim of this study is to determine whether antibiotic treatment could reduce mechanical ventilation duration in patients with nosocomial tracheobronchitis acquired under mechanical ventilation.

DETAILED DESCRIPTION:
Rationale:

Ventilator-associated tracheobronchitis (VAT) is common in intensive care unit (ICU) patients, rates of 2.7%-10.6% are reported in the literature. This nosocomial infection is associated with weaning difficulties resulting in prolonged duration of mechanical ventilation (MV) and ICU stay. A case-control study performed in chronic obstructive pulmonary disease (COPD) patients with VAT found antibiotic treatment to be significantly associated with reduced duration of MV. Another case control-study, performed in VAT patients without chronic respiratory failure, found no significant difference in duration of MV between patients who received adequate antibiotic treatment and those who received inadequate antibiotic treatment. In addition, antibiotic use is known to be associated with subsequent multidrug-resistant bacteria (MRB), longer duration of MV, and mortality rates. Therefore, a randomized controlled study is necessary to determine the impact of antibiotic treatment on outcome in VAT patients.

Patients and methods:

390 patients will be included in this prospective randomized open multicenter study. Inclusion of 390 patients is required to demonstrate a significant reduction of MV duration of 5 days (α = 0.025, β = 0.10). An intermediate analysis will be performed. All patients intubated and ventilated > 48h who developed a first episode of VAT are eligible. Primary endpoint is the duration of MV. Secondary end points are ICU length of stay, mortality, ventilator-associated pneumonia, ICU-acquired infection, MRB, and yeast rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tracheobronchitis diagnosed after 48h of invasive mechanical ventilation

Exclusion Criteria:

* Immunodepressed patients
* Patients with tracheostomy at ICU admission
* Patients who developed ventilator-associated pneumonia before ventilator-associated tracheobronchitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-06; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
duration of mechanical ventilation

SECONDARY OUTCOMES:
length of intensive care unit (ICU) stay
mortality rate
ventilator-associated pneumonia rate

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD, Principal Investigator — University Hospital of Lille
Locations (1):
- 12 ICUs in north of France, Lille, France

REFERENCES:
- [Derived] Nseir S, Favory R, Jozefowicz E, Decamps F, Dewavrin F, Brunin G, Di Pompeo C, Mathieu D, Durocher A; VAT Study Group. Antimicrobial treatment for ventilator-associated tracheobronchitis: a randomized, controlled, multicenter study. Crit Care. 2008;12(3):R62. doi: 10.1186/cc6890. Epub 2008 May 2. PMID 18454864